CLINICAL TRIAL: NCT07347626
Title: Efficacy and Safety of Eptifibatide Therapy Following Intravenous Thrombolysis in Acute Ischemic Stroke Patients Within 4.5 to 24 Hours After Onset: A Multicenter, Randomized Controlled Trial
Brief Title: Eptifibatide for Extended Window Ischemic Stroke After Thrombolysis
Acronym: E-TWIST
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: The First Affiliated Hospital of Hainan Medical College (Unknown); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-TWIST
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Intravenous thrombolysis; Eptifibatide; Neurological deterioration
MeSH Terms: conditions — Ischemic Stroke | interventions — Eptifibatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eptifibatide (Integrilin) (Experimental): Participants randomized to this arm will receive intravenous eptifibatide (135 μg/kg bolus, followed by 0.75 μg/kg/min infusion for 2 hours) initiated within 60 minutes after completion of standard intravenous thrombolysis (either alteplase or tenecteplase). Antiplatelet therapy with aspirin (100 mg) and/or clopidogrel (75 mg) will be administered at 24h after thrombolysis until the follow-up period of 90 days.
  Interventions: Drug: Eptifibatide (Integrilin)
- Standard Medical Therapy (Active Comparator): Participants randomized to this arm will not receive intravenous eptifibatide after completion of standard intravenous thrombolysis. Antiplatelet therapy with aspirin (100 mg) and/or clopidogrel (75 mg) will be administered at 24h after thrombolysis until the follow-up period of 90 days.
  Interventions: Drug: Standard Medical Therapy

INTERVENTIONS:
Drug: Eptifibatide (Integrilin) — Participants will receive intravenous eptifibatide (135 μg/kg bolus, followed by 0.75 μg/kg/min infusion for 2 hours) initiated within 60 minutes after completion of standard intravenous thrombolysis (either alteplase or tenecteplase). Antiplatelet therapy with aspirin (100 mg) and/or clopidogrel (75 mg) will be administered at 24h after thrombolysis until the follow-up period of 90 days.
  Arms: Eptifibatide (Integrilin)
Drug: Standard Medical Therapy — Participants will not receive intravenous eptifibatide after completion of standard intravenous thrombolysis. Antiplatelet therapy with aspirin (100 mg) and/or clopidogrel (75 mg) will be administered at 24h after thrombolysis until the follow-up period of 90 days.
  Arms: Standard Medical Therapy

SUMMARY:
This is a multicenter, randomized, open-label, blinded-endpoint clinical trial designed to evaluate the efficacy and safety of early administration of eptifibatide following intravenous thrombolysis in patients with acute ischemic stroke who present 4.5 to 24 hours after symptom onset.

DETAILED DESCRIPTION:
Several clinical trials (e.g., TRACE-3, EXPECTS, HOPE) have successfully extended the time window for intravenous thrombolysis (IVT) from the conventional 4.5 hours up to 24 hours after symptom onset by utilizing advanced imaging selection techniques. Consequently, the 2024 Chinese guidelines for reperfusion therapy recommend IVT for patients presenting 4.5 to 24 hours after onset, based on imaging selection criteria. However, clinical practice indicates that a considerable proportion of patients exhibit suboptimal recanalization outcomes or even experience early neurological deterioration (END) despite receiving standard IVT. Previous research, such as the ASSET-IT trial, has primarily focused on patients treated within 4.5 hours of onset. For the growing population of "extended-window" (4.5-24 hours) patients receiving IVT facilitated by advances in imaging, the optimal antiplatelet strategy following thrombolysis remains an area with no high-level evidence. Therefore, this study aims to evaluate the efficacy and safety of early administration of eptifibatide following standard IVT (with tenecteplase or alteplase) in patients with acute ischemic stroke who present 4.5 to 24 hours after symptom onset. Patients who have received standard IVT but exhibit early neurological deterioration, fluctuation, or lack of significant improvement within 1 hour post-thrombolysis will be randomized 1:1 to receive either eptifibatide (a single intravenous bolus followed by a 2-hour infusion) plus standard medical therapy or standard medical therapy alone. The primary efficacy outcome is the proportion of patients achieving an excellent functional outcome (modified Rankin Scale score of 0-1) at 90 days. The primary safety outcome is the incidence of symptomatic intracranial hemorrhage within 48 hours after randomization. A total of 786 participants are planned to be enrolled to detect a 10% absolute difference in the primary outcome with 80% power.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Acute ischemic stroke, with the time interval from last known well to hospital presentation being 4.5 to 24 hours.
3. NIHSS score ≥ 4 before randomization; if large or medium vessel occlusion is present, an NIHSS score ≤ 10 is also required.
4. Presence of any of the following conditions after completion of standard intravenous thrombolysis:

   1. No significant neurological improvement within 1 hour (defined as a change in NIHSS score ≤ 1 point from baseline).
   2. Early neurological deterioration within 1 hour of onset (defined as an increase in NIHSS score ≥ 2 points from baseline).
   3. Neurological fluctuation within 24 hours after symptom onset (defined as an increase in NIHSS score ≥ 2 points from the lowest value post-thrombolysis).
5. Ability to receive the assigned study drug within 60 minutes after intravenous thrombolysis.
6. Signed written informed consent obtained from the patient or their legal representative.

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by CT or MRI.
2. Planned endovascular therapy.
3. Presence of any definite cardioembolic source, including: chronic or paroxysmal atrial fibrillation, sick sinus syndrome, mitral stenosis, mechanical heart valve, endocarditis, intracardiac thrombus or vegetation, myocardial infarction within 3 months, dilated cardiomyopathy, spontaneous echo contrast in the left atrium, or ejection fraction < 30%.
4. Pre-stroke modified Rankin Scale (mRS) score ≥ 2.
5. Renal insufficiency (glomerular filtration rate < 30 ml/min or serum creatinine > 220 μmol/L [2.5 mg/dL]).
6. Known hypercoagulable state.
7. Platelet count < 100 × 10⁹/L.
8. Pregnancy or lactation.
9. Allergy to eptifibatide, other glycoprotein IIb/IIIa inhibitors, aspirin, or clopidogrel.
10. History of non-atherosclerotic arteriopathy, including moyamoya disease, arterial dissection, or fibromuscular dysplasia.
11. Pre-existing neurological or psychiatric disease that would preclude accurate neurological assessment.
12. History of bleeding diathesis, severe cardiac disease, liver disease, or sepsis.
13. Brain tumor with mass effect on imaging (except for small meningiomas).
14. Evidence of intracranial arteriovenous malformation or aneurysm with diameter > 5 mm on CT or MR angiography.
15. Current participation in another clinical trial.
16. Any terminal illness with life expectancy < 6 months.
17. Anticipated inability to complete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Excellent functional outcome | 90 days post-randomization
  modified Rankin scale score of 0 to 1. modified Rankin scale scores range from 0 to 6, with 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.

SECONDARY OUTCOMES:
Ordinal degree of disability | 90 days post-randomization
  Ordinal degree of disability on the modified Rankin scale score at 90 days (shift analysis)
Conversion to Endovascular Therapy | 24 hours post-randomization
  Proportion of patients who converted to endovascular therapy
Functionally independent | 90 days post-randomization
  modified Rankin scale score of 0 to 2
Change in NIHSS Score at 48 (±12) Hours | 48 (±12) hours post-randomization
  Change in NIHSS score from pre-randomization to 48 (±12) hours
Change in NIHSS Score at Discharge or Day 6 (±1) | Day 6 (±1) or discharge post-randomization, whichever came first
  Change in NIHSS score from pre-randomization to discharge or day 6 (±1)
Health-related quality of life | 90 days post-randomization
  assessed with the European Quality Five Dimensions Five Level scale
Symptomatic intracranial hemorrhage | 48 (±12) hours post-randomization
  defined as per the Heidelberg bleeding classification
Mortality | 90 days post-randomization
  The proportion of participants who die from any cause within 90 days after randomization in the study
Incidence of major extracranial bleeding within 48 (±12) hours | 48 (±12) hours post-randomization
  GUSTO criteria: moderate and severe bleeding
Incidence of non-hemorrhagic serious adverse events | Within 90 days post-randomization
  Including but not limited to cerebral herniation, pneumonia, respiratory failure, circulatory failure, stress ulcer, secondary epilepsy, urinary tract infection, sepsis, renal failure, acute coronary syndrome, venous thrombosis, and psychiatric symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Zhongming Qiu, MD, Principal Investigator — Xinqiao Hospital of the Army Medical University; Zhenqiang Zhao, MD, Principal Investigator — The First Affiliated Hospital of Hainan Medical University; Daojun Hong, MD, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (6):
- China (6):
  - Xinqiao Hospital and The Second Affiliated Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The Affiliated Hospital of Jinggangshan University, Ji’an, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bonita R, Beaglehole R. Recovery of motor function after stroke. Stroke. 1988 Dec;19(12):1497-500. doi: 10.1161/01.str.19.12.1497. PMID 3201508
- [Result] Seners P, Ben Hassen W, Lapergue B, Arquizan C, Heldner MR, Henon H, Perrin C, Strambo D, Cottier JP, Sablot D, Girard Buttaz I, Tamazyan R, Preterre C, Agius P, Laksiri N, Mechtouff L, Bejot Y, Duong DL, Mounier-Vehier F, Mione G, Rosso C, Lucas L, Papassin J, Aignatoaie A, Triquenot A, Carrera E, Niclot P, Obadia A, Lyoubi A, Garnier P, Crainic N, Wolff V, Tracol C, Philippeau F, Lamy C, Soize S, Baron JC, Turc G; MINOR-STROKE Collaborators. Prediction of Early Neurological Deterioration in Individuals With Minor Stroke and Large Vessel Occlusion Intended for Intravenous Thrombolysis Alone. JAMA Neurol. 2021 Mar 1;78(3):321-328. doi: 10.1001/jamaneurol.2020.4557. PMID 33427887
- [Result] Han L, Hou Z, Ma M, Ding D, Wang D, Fang Q. Impact of glycosylated hemoglobin on early neurological deterioration in acute mild ischemic stroke patients treated with intravenous thrombolysis. Front Aging Neurosci. 2023 Jan 12;14:1073267. doi: 10.3389/fnagi.2022.1073267. eCollection 2022. PMID 36711206
- [Result] Yang T, Fan K, Cao Y, Yan J, Han Z. Stroke Type, Etiology, Clinical Features and Prognosis of Diabetic Patients in Southern China. Clin Appl Thromb Hemost. 2020 Jan-Dec;26:1076029620973090. doi: 10.1177/1076029620973090. PMID 33296224
- [Result] Tu WJ, Chao BH, Ma L, Yan F, Cao L, Qiu H, Ji XM, Wang LD. Case-fatality, disability and recurrence rates after first-ever stroke: A study from bigdata observatory platform for stroke of China. Brain Res Bull. 2021 Oct;175:130-135. doi: 10.1016/j.brainresbull.2021.07.020. Epub 2021 Jul 27. PMID 34329730
- [Result] Wang M, Wang CJ, Gu HQ, Meng X, Jiang Y, Yang X, Zhang J, Xiong YY, Zhao XQ, Liu LP, Wang YL, Wang YJ, Li ZX. Sex Differences in Short-Term and Long-Term Outcomes Among Patients With Acute Ischemic Stroke in China. Stroke. 2022 Jul;53(7):2268-2275. doi: 10.1161/STROKEAHA.121.037121. Epub 2022 Feb 8. PMID 35130717
- [Result] Wang W, Jiang B, Sun H, Ru X, Sun D, Wang L, Wang L, Jiang Y, Li Y, Wang Y, Chen Z, Wu S, Zhang Y, Wang D, Wang Y, Feigin VL; NESS-China Investigators. Prevalence, Incidence, and Mortality of Stroke in China: Results from a Nationwide Population-Based Survey of 480 687 Adults. Circulation. 2017 Feb 21;135(8):759-771. doi: 10.1161/CIRCULATIONAHA.116.025250. Epub 2017 Jan 4. PMID 28052979
- [Result] The Lancet Public Health. Strengthening public health for a Healthy China. Lancet Public Health. 2021 Dec;6(12):e866. doi: 10.1016/S2468-2667(21)00261-9. No abstract available. PMID 34838189